CLINICAL TRIAL: NCT05788406
Title: Does Dynamic Balance Exercises Affect Flexible Pes Planus?
Brief Title: Effects of Dynamic Balance Exercise on Flexible Pes Planus
Acronym: PesPlanus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Eylül Pınar KISA, Lecturer, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BirUni
Record Dates: First submitted 2023-03-14; First posted 2023-03-28 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Pes Planus
Keywords: flexible pes planus; insole; balance
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short Foot Exercises Group (Experimental): İnsole+Short Foot Exercises group
  Interventions: Other: Short foot exercises, Dynamic balance exercises and insole
- Balance Exercises Group (Experimental): İnsole+Balance exercises group
  Interventions: Other: Short foot exercises, Dynamic balance exercises and insole
- Control Group (Experimental): İnsole group
  Interventions: Other: Short foot exercises, Dynamic balance exercises and insole

INTERVENTIONS:
Other: Short foot exercises, Dynamic balance exercises and insole — Short foot exercises is used to improve muscle strenght, Dynamic balance exercises is used to improve balance and insole is used to improve MLA

SUMMARY:
The purpose of this study is to investigate the effects of intrinsic strengthening and dynamic balance exercises in patients with flexible pes planus. Forty-five participants aged 18 to 35 years were enrolled in the study, and the first group underwent intrinsic foot muscle strengthening training with short foot exercises (SFE) and used insoles. The second group trained using the dynamic balance board, which promotes dynamic balance and used insoles. The third group used only insoles. The total duration of treatment was 8 weeks/3 days. The degree of foot deformity was assessed with the, medial longitudinal arch (MLA) angle, measurements of subtalar angle and navicular drop test. Foot position assessed using Foot Posture Index (FPI) Static balance was assessed with the Flamingo Balance Test and dynamic balance with the " BOBO Health Platform with Gaming®" device.

DETAILED DESCRIPTION:
Pes planus (flatfoot) is generally defined as valgus of the hindfoot, disappearance of the medial longitudinal arch (MLA) in the midfoot, and supination of the forefoot relative to the hindfoot when the foot is loaded. MLA height is the most important measurement for determining the degree of pes planus. The decrease in MLA disrupts this balance and causes the muscles and bones that are supposed to balance the effect of external forces to be subjected to greater stress. As a result, the balance is affected. Conservative treatment options that can be used as the first step in treating pes planus include activity modifications, exercises, manipulations, serial cast applications, weight loss, shoes changes, shoes modifications, use of foot orthotics. Several methods are used to strengthen foot intrinsic muscles, including toe towel curls, picking up objects, shin curls, unilateral balance activities, and the short foot exercise. The common exercises are strengthening exercises defined for intrinsic muscles, "short foot exercises" (SF). It is known that arch support insoles improve foot malalignment, correct dynamic posture, effectively support leg alignment and pain relief, and normalize gait. The use of silicone insoles is a product whose range of application has increased in recent years. The extremely soft and flexible material ensures that the shape of the foot is adopted. The researchers believed that the presence of a pes planus foot deformity, common in young people, negatively affects the balance of the individual, revealing small disturbances and different balance strategies. In this situation, the training of intrinsic muscles is of great importance. The investigators aim in this study is to investigate the effects of intrinsic muscle strengthening and dynamic balance exercises performed with silicone soles in individuals with flexible pes planus.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included in the study if they were 152° above the MLA, participants with flexible pes planus at the 1st, 2nd, and 3rd level according to Jack's test, between 18 and 35 years of age, and had not received previous treatment for pes planus.

Exclusion Criteria:

* Individuals who had previously used orthotics, who had an orthopedic injury to the ankle, and who did not wish to participate in the study were excluded from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Dynamic Balance performance | 0-8 week
  Dynamic balance was assessed using the BOBO Gaming Health Platform. With this system, which acts as a computerized strength platform, there are assessment and treatment phases. The individual was performed with the foot being tested on 2 sides of the platform. In all these evaluations, parameters related to body balance were analyzed. It gives performance scores in terms of percent.

SECONDARY OUTCOMES:
Foot Posture Index Score | 0-8 week
  Foot posture was analyzed using the Foot Posture Index. Palpation of the head of the talus in the hindfoot, inclination below and above the lateral malleolus, pronation/supination of the calcaneus, ballooning at the talonavicular joint in the forefoot, MLA structure, and abduction/adduction of the forefoot relative to the hindfoot were evaluated. Each of these criteria was assigned scores ranging from -2 to +2. The total score obtained was recorded and it indicated that the foot was in neutral position at 0, in pronation at positive values and in supination at negative values.
Subtalar angle | 0-8 week
  Measurement of the subtalar angle between the Achilles tendon and the midpoint of the calcaneus was measured while the patient stood on a high platform. The pivot point was assumed to be 1 cm below the medial malleolus, and this area was marked. An angle greater than 5 degrees in the pronation or supination direction was considered abnormal.
Static Balance Assessment | 0-8 week
  The patient flexed the foot behind the knee and held it with the hand in the same direction. When the patient was ready, he released the hand of the physiotherapist and at the same time the stopwatch was started. Each time the patient lost balance (touching the floor, releasing the foot), the stopwatch was stopped and restarted when the patient was ready 60 seconds. The total number of balance losses during this period was reported with number
Angle of Medial longitudinal Arch | 0-8 week
  While measuring the MLA angle, a line was drawn from the center of the medial malleolus to the center of the navicular. The other line was drawn from the tuberosity of the navicular to the center of the first metatarsal head. The angle between these two lines was measured with a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: EylÜL pINAR Kısa, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)